CLINICAL TRIAL: NCT03313193
Title: Acupressure Intervention to Reduce Treatment-related Symptoms in Children With Cancer or Receiving a Hematopoietic Stem Cell Transplant
Brief Title: Acupressure for Children in Treatment for a Childhood Cancer
Acronym: ACT-CC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Pierre's Birthday Fund (Unknown)
Responsible Party: Principal Investigator, Anne Lown, E. Anne Lown, Dr.P.H., Associate Adjunct Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 170820
Record Dates: First submitted 2017-08-22; First posted 2017-10-18 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Treatment-Related Cancer
Keywords: nausea; vomiting; pain; fatigue; depression; anxiety; PTSD-parent; caregiver self efficacy-parent
MeSH Terms: conditions — Neoplasms, Second Primary; Nausea; Vomiting; Pain; Fatigue; Depression; Anxiety Disorders | interventions — Acupressure; Therapeutics

STUDY DESIGN:
Intervention Model Description: Pragmatic Randomized Controlled Trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Acupressure for Children in Treatment for a Childhood Cancer + usual care
  Interventions: Other: Acupressure for Children in Treatment for a Childhood Cancer
- Arm B (No Intervention): Usual care alone

INTERVENTIONS:
Other: Acupressure for Children in Treatment for a Childhood Cancer — This study will describe the benefits and risks of an acupressure intervention to decrease nausea/vomiting and other treatment-related symptoms compared to a control group receiving usual care. Children in Arm A will receive usual symptom management care + acupressure 5 days/week for ~20 treatments. Parents will be taught how to provide acupressure as well. Children in Arm B will receive usual care alone.
  Arms: Arm A

SUMMARY:
Background: Despite advances in symptom management, children undergoing cancer treatment or receiving a chemotherapy-based Hematopoietic Stem Cell Transplant (HSCT) often suffer from moderate to severe symptoms of nausea/vomiting, pain, and fatigue along with psychological distress. Pharmacologic treatments of symptoms can cause side-effects. Patients, parents, and clinicians have expressed interest in including non-pharmacologic approaches to improve symptom management. Acupuncture/acupressure is a promising adjunctive therapy to usual care. More evidence is needed from well-designed trials with larger samples and rigorous designs in order to make definitive recommendations about the routine inclusion of acupressure among pediatric patients being treated for childhood cancer or receiving a HSCT.

Design and Methods 100 dyads (one child with one parent/caregiver) will be randomized 1:1 into 2 study arms (50 children in each arm). Arm A participants will be offered usual care and professional acupressure five times weekly (15-20 minute sessions) and a parent/caregiver will be instructed in acupressure delivery for the child as symptoms arise. Arm B participants will receive usual care alone. (At the study end, Arm B parents will be offered acupressure instructions.) Children will be enrolled for ~30 days which can occur with one month of continuous hospital-based treatment or two months of intermittent hospital-based treatment (inpatient or regular outpatient treatment). Parent and child participants will receive a follow-up interview one month after completion of the intervention (Arm A) or the final symptom assessment (Arm B).

Significance This is the first study to evaluate the effectiveness and safety of an acupressure intervention to decrease treatment-related symptoms in 100 patients in treatment for a childhood cancer or receiving a chemo-therapy based HSCT.

DETAILED DESCRIPTION:
AIMS

Aim 1: To assess the feasibility of an acupressure intervention plus usual care and to assess the benefits and risks compared to usual care alone for children receiving hospital-based treatment for a childhood cancer or a HSCT. The study hypothesizes that patients in the acupressure arm will report decreased nausea/vomiting and improved management of treatment -related symptoms compared to the usual care only arm. We will test the following hypotheses:

1a. Primary outcomes: Children receiving acupressure will report reduced nausea/vomiting measured as a composite variable compared to the usual care alone group.

1b. Secondary outcomes: Children receiving the acupressure intervention will have reduced levels of each; nausea, vomiting, and rescue antiemetic use compared to the usual care alone group.

1c. Secondary outcomes: Children receiving acupressure will report reduced pain interference and pain intensity, reduced fatigue, anxiety, depression, other treatment-related symptoms, and greater positive affect compared to the usual care group. Children receiving acupressure will use less rescue pain medication compared to the usual care alone group.

1. d. Greater dose of acupressure will lead to greater improvement of primary and secondary outcomes.

   Aim 2: To assess the benefits and challenges of providing the acupressure intervention for parents.
2. a. The parent/caregiver in Arm A will report decreased post-traumatic stress symptoms, reduced anxiety and depression, and increased caregiving self-efficacy 4 weeks after the end of professional acupressure. 2b. An open-ended question for parents/caregivers in the intervention arm will elicit information on the experience of providing acupressure for their children.

Additional Qualitative Aims:

Qualitative Aim 1: To explore the child's experience of receiving acupressure and the caregiver's experience of delivering acupressure to the child through a semi-structured interview with the caregiver, with a focus on well-being. We will explore how acupressure impacts the proposed components of well- being: hedonistic and eudemonic perspectives of positive feelings, as well as the less studied somatic and physical components such as mind-body integration and increased connection through touch in the child and caregiver.

Qualitative Aim 2: To explore the acupressure provider's impression of how provider- or caregiver- delivered acupressure impacts the child's experience of childhood cancer treatment or HSCT.

DESIGN The goal of the study is to describe the benefits and risks of an acupressure intervention to decrease nausea/vomiting and other treatment-related symptoms compared to a control group receiving usual care. This study is a pragmatic randomized clinical trial. Participants will be randomized 1:1 into 2 study arms. In Arm A children will be offered professional acupressure five times weekly along with usual care for ~30 days of hospital-based treatment (continuous in-hospital) or two months of hospital-based treatment (intermittent) for an approximate total of 20 semi-standardized acupressure treatments. Treatments take approximately 20 minutes each. A parent/caregiver will be instructed in how to deliver acupressure to his/her child as symptoms arise using a simplified protocol with supplemental educational handouts. In Arm B participants will receive usual care alone. All usual care is defined according to COG supportive care guidelines. After the final study assessment parents/caregivers will be given instruction on how to deliver acupressure. Outcomes will be assessed in all children in Arm A and Arm B at baseline, 5 days a week for nausea, vomiting, and pain, two times a week for remaining symptoms, and at a once month follow-up. Outcomes will be assessed in caregivers at baseline, ~day 7, and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Children who are either receiving treatment for diagnosis of a childhood cancer (curative or supportive care) or are receiving a chemotherapy-based HSCT. Non-malignant brain central nervous system tumors are considered as a childhood cancer.
2. Ages 5- 24 years old.
3. Be receiving hospital-based treatment (inpatient or outpatient) so that acupressure treatments can be delivered and parents can be trained and monitored.
4. Availability and willingness of a parent or caregiver to deliver acupressure for ages 5-17. For young adults ages 18-24 participation of a parent, close friend or family member/caregiver is preferred but not required.
5. English or Spanish speaking.
6. Receiving treatment at UCSF Benioff Children's Hospital.

Exclusion Criteria

1) Children/young adults who meet the above criteria, but whose treating oncologist, health care provider, or a study investigator advises against study participation for physical health, mental health (parent or child) or logistical reasons.

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Decrease in nausea/vomiting severity | past 24 hours for nausea/vomiting measures daily over 30 days of hospital-based treatment (continuous hospitalization or intermittent treatment over 2 months)
  assessed using the Pediatric Nausea Assessment Tool (PeNAT)(Dupuis, 2006)(see description below) + a single Question on vomiting for ages 5-17. The MASCC Anti-emesis Tool (MAT) will be used to assess nausea (yes/no) and severity for ages 18+.This composite measure of nausea/vomiting in the child represents a continuum of nausea/vomiting (range=1-8).

SECONDARY OUTCOMES:
Decreased nausea (PeNAT) | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  Nausea will be measured using the PeNat scale, validated for ages 4-17 years. Four levels of nausea are defined on this scale: none, mild, moderate and severe, using faces, a preferred method of measuring distress among children. In the case where a child cannot report on nausea, parent report will be sought. Parents report of child's nausea severity was found to be significantly correlated with child reports. Patients ages 18-24 will be given the MAT.
Decreased vomiting (Vol, 2016) | 30 days hospitalization (continuous or intermittent over 2 months)
  Vomiting episodes will be measured as recorded by patients and families using patient diaries (confirmed using review of daily patient electronic medical records (EMR)). Vomiting episodes will be capped so the range will be 1-4+ episodes in the 2 day time-span since the last assessment. Using these two variables we can construct a variable for no nausea and no vomiting which is typically called "complete control" and is a standard outcome for many pharmaceutical antiemetic trials.
Use of fewer rescue anti-emetics (from Electronic Medical Records) | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  This will be categorized as a 1-4+ variable where 1=no rescue antiemetic use and 4+ means that a dose was taken 4 or more times between assessments. (Emetogenicity will be assessed using the newest guidelines.) From electronic medical records (EMR).
Complete control of nausea/vomiting | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  Using the nausea and vomiting variables we will construct a dichotomous variable for no nausea and no vomiting which is typically called "complete control" and is a standard outcome for many pharmaceutical antiemetic trials.
Decreased pain interference assessed using the PROMIS Pediatric Pain Interference Scale | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  (4 items) from the Pediatric Profile 25 v. 2. Pediatric or Parent Proxy Versions assess pain interference in the context of daily activities including interference on physical, psychological and social functioning. (Varni, 2010)
Decreased Pain intensity | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  PROMIS Pediatric or Parent Proxy Version includes 1 question that assesses intensity of pain on a 0-10 scale. This single-item pain intensity question is included in the Pediatric Profile 25 v2 and is not scored but reported using a raw score (e.g., 0 to 10).
Decreased pain assessed (ages 5-7) | 30 days of hospital-based treatment (continuous or intermittent over 2 months)
  Faces Pain (Intensity) Scale-Revised (FPS-R)(1 item) children rank severity of pain using 6 gender-neutral faces depicting 'no pain' to 'most pain'; scores range from 0 to 10.
Decreased fatigue symptoms | 30 days of hospital-based treatment (continuous or intermittent over 2 months)
  PROMIS Pediatric Profile 25 v2. This 4-item scale includes two domains: feeling tired and (lack of) energy and its impact on daily life.
Decreased depression symptoms | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  (4 items) from PROMIS pediatric profile 25 v 2.0 Among young adults aged 18+. 4-item subscales of PROMIS Adult Profile 29 v2.0 will be used.
Decreased anxiety | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  (4 items) from PROMIS pediatric profile 25 v 2.0
Increased Well-being | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  PROMIS Pediatric Positive Affect measure. This measures positive emotions (well-being) which can reduce experience of symptom burden and protect health. (4 items) Among parents/caregivers the study used Positive Affect Subscale of the PANAS (5-items): This positive affect sub-scale of the 10-item PANAS scale (i-PANAS-SF) assesses positive or pleasurable engagement with the environment, well-being, and satisfaction with life.
Fewer overall symptoms assessed using the Symptom Screening in Pediatrics (SSPedi) tool (Tomlinson, 2014) | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  This pediatric cancer-specific symptom screening and assessment scale measures physical and psychological symptoms (e.g., feeling angry, sad or worried, tired, mouth sores, headache, constipation or diarrhea, problems thinking or remembering, body changes, or appetite loss, among others) in 15 questions.
Decreased depression symptoms using the PROMIS depression (adult) measure. | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  4 item measure used to assess depression among the child's parent/caregiver using subscales of PROMIS Adult Profile 29 v2.0 will be used.
Decreased anxiety assessed using PROMIS anxiety (adult) | 30 days hospital-based treatment (continuous or intermittent over 2 months)
  4 item measure used to assess anxiety among the child's parent/caregiver using subscales of PROMIS Adult Profile 29 v2.0 will be used.
Fewer PTSD symptoms, (PCL-5) (adult) | 1 month after end of 30 days trial enrollment
  the Post-traumatic Stress Disorder Checklist is a 20 item measure - updated to use DSM5 criteria. Responses assess frequency and intensity of symptoms (strong internal consistency, test-retest reliability and validity). Total symptom scores will be compared between groups.
Increased Caregiver Self-Efficacy (parent) | 1 month after end of 30 day trial enrollment
  This 6 item scale is adapted from Bandura, 1977, Lorig, 1989; Barlow, 2000) and previously used in parents of children with disabilities (excellent psychometric reliability and validity).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lown, Dr.P.H., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Background] Roscoe JA, Morrow GR, Hickok JT, Bushunow P, Pierce HI, Flynn PJ, Kirshner JJ, Moore DF, Atkins JN. The efficacy of acupressure and acustimulation wrist bands for the relief of chemotherapy-induced nausea and vomiting. A University of Rochester Cancer Center Community Clinical Oncology Program multicenter study. J Pain Symptom Manage. 2003 Aug;26(2):731-42. doi: 10.1016/s0885-3924(03)00254-9. PMID 12906958
- [Background] Mao JJ, Xie SX, Bowman MA. Uncovering the expectancy effect: the validation of the acupuncture expectancy scale. Altern Ther Health Med. 2010 Nov-Dec;16(6):22-7. PMID 21280459
- [Background] Forrest CB, Bevans KB, Tucker C, Riley AW, Ravens-Sieberer U, Gardner W, Pajer K. Commentary: the patient-reported outcome measurement information system (PROMIS(R)) for children and youth: application to pediatric psychology. J Pediatr Psychol. 2012 Jul;37(6):614-21. doi: 10.1093/jpepsy/jss038. Epub 2012 Feb 23. No abstract available. PMID 22362923
- [Background] Garcia SF, Cella D, Clauser SB, Flynn KE, Lad T, Lai JS, Reeve BB, Smith AW, Stone AA, Weinfurt K. Standardizing patient-reported outcomes assessment in cancer clinical trials: a patient-reported outcomes measurement information system initiative. J Clin Oncol. 2007 Nov 10;25(32):5106-12. doi: 10.1200/JCO.2007.12.2341. PMID 17991929
- [Background] DeWitt EM, Stucky BD, Thissen D, Irwin DE, Langer M, Varni JW, Lai JS, Yeatts KB, Dewalt DA. Construction of the eight-item patient-reported outcomes measurement information system pediatric physical function scales: built using item response theory. J Clin Epidemiol. 2011 Jul;64(7):794-804. doi: 10.1016/j.jclinepi.2010.10.012. Epub 2011 Feb 2. PMID 21292444
- [Background] Irwin DE, Stucky B, Langer MM, Thissen D, Dewitt EM, Lai JS, Varni JW, Yeatts K, DeWalt DA. An item response analysis of the pediatric PROMIS anxiety and depressive symptoms scales. Qual Life Res. 2010 May;19(4):595-607. doi: 10.1007/s11136-010-9619-3. Epub 2010 Mar 7. PMID 20213516
- [Background] Varni JW, Stucky BD, Thissen D, Dewitt EM, Irwin DE, Lai JS, Yeatts K, Dewalt DA. PROMIS Pediatric Pain Interference Scale: an item response theory analysis of the pediatric pain item bank. J Pain. 2010 Nov;11(11):1109-19. doi: 10.1016/j.jpain.2010.02.005. Epub 2010 Jun 2. PMID 20627819
- [Background] Kashikar-Zuck S, Carle A, Barnett K, Goldschneider KR, Sherry DD, Mara CA, Cunningham N, Farrell J, Tress J, DeWitt EM. Longitudinal evaluation of patient-reported outcomes measurement information systems measures in pediatric chronic pain. Pain. 2016 Feb;157(2):339-347. doi: 10.1097/j.pain.0000000000000378. PMID 26447704
- [Background] Varni JW, Thissen D, Stucky BD, Liu Y, Gorder H, Irwin DE, DeWitt EM, Lai JS, Amtmann D, DeWalt DA. PROMIS(R) Parent Proxy Report Scales: an item response theory analysis of the parent proxy report item banks. Qual Life Res. 2012 Sep;21(7):1223-40. doi: 10.1007/s11136-011-0025-2. Epub 2011 Oct 5. PMID 21971875
- [Background] Irwin DE, Gross HE, Stucky BD, Thissen D, DeWitt EM, Lai JS, Amtmann D, Khastou L, Varni JW, DeWalt DA. Development of six PROMIS pediatrics proxy-report item banks. Health Qual Life Outcomes. 2012 Feb 22;10:22. doi: 10.1186/1477-7525-10-22. PMID 22357192
- [Background] Hinds PS, Nuss SL, Ruccione KS, Withycombe JS, Jacobs S, DeLuca H, Faulkner C, Liu Y, Cheng YI, Gross HE, Wang J, DeWalt DA. PROMIS pediatric measures in pediatric oncology: valid and clinically feasible indicators of patient-reported outcomes. Pediatr Blood Cancer. 2013 Mar;60(3):402-8. doi: 10.1002/pbc.24233. Epub 2012 Jul 24. PMID 22829446
- [Background] Lai JS, Stucky BD, Thissen D, Varni JW, DeWitt EM, Irwin DE, Yeatts KB, DeWalt DA. Development and psychometric properties of the PROMIS((R)) pediatric fatigue item banks. Qual Life Res. 2013 Nov;22(9):2417-27. doi: 10.1007/s11136-013-0357-1. Epub 2013 Feb 2. PMID 23378106
- [Background] Vol H, Flank J, Lavoratore SR, Nathan PC, Taylor T, Zelunka E, Maloney AM, Lee Dupuis L. Poor chemotherapy-induced nausea and vomiting control in children receiving intermediate or high dose methotrexate. Support Care Cancer. 2016 Mar;24(3):1365-71. doi: 10.1007/s00520-015-2924-1. Epub 2015 Sep 3. PMID 26335406
- [Background] Dupuis LL, Taddio A, Kerr EN, Kelly A, MacKeigan L. Development and validation of the pediatric nausea assessment tool for use in children receiving antineoplastic agents. Pharmacotherapy. 2006 Sep;26(9):1221-31. doi: 10.1592/phco.26.9.1221. PMID 16945043
- [Background] Dupuis LL. Chemotherapy-induced vomiting in children: some progress, more questions. Lancet Oncol. 2016 Mar;17(3):264-265. doi: 10.1016/S1470-2045(15)00582-3. Epub 2016 Jan 19. No abstract available. PMID 26795845
- [Background] Bieri D, Reeve RA, Champion DG, Addicoat L, Ziegler JB. The Faces Pain Scale for the self-assessment of the severity of pain experienced by children: development, initial validation, and preliminary investigation for ratio scale properties. Pain. 1990 May;41(2):139-150. doi: 10.1016/0304-3959(90)90018-9. PMID 2367140
- [Background] Stinson JN, Kavanagh T, Yamada J, Gill N, Stevens B. Systematic review of the psychometric properties, interpretability and feasibility of self-report pain intensity measures for use in clinical trials in children and adolescents. Pain. 2006 Nov;125(1-2):143-57. doi: 10.1016/j.pain.2006.05.006. Epub 2006 Jun 13. PMID 16777328
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Tsze DS, Hirschfeld G, von Baeyer CL, Bulloch B, Dayan PS. Clinically significant differences in acute pain measured on self-report pain scales in children. Acad Emerg Med. 2015 Apr;22(4):415-22. doi: 10.1111/acem.12620. Epub 2015 Mar 13. PMID 25773461
- [Background] Powell CV, Kelly AM, Williams A. Determining the minimum clinically significant difference in visual analog pain score for children. Ann Emerg Med. 2001 Jan;37(1):28-31. doi: 10.1067/mem.2001.111517. PMID 11145767
- [Background] O'Sullivan C, Dupuis LL, Gibson P, Johnston DL, Baggott C, Portwine C, Spiegler B, Kuczynski S, Tomlinson D, de Mol Van Otterloo S, Tomlinson GA, Sung L. Refinement of the symptom screening in pediatrics tool (SSPedi). Br J Cancer. 2014 Sep 23;111(7):1262-8. doi: 10.1038/bjc.2014.445. Epub 2014 Aug 7. PMID 25101569
- [Background] Tomlinson D, Dupuis LL, Gibson P, Johnston DL, Portwine C, Baggott C, Zupanec S, Watson J, Spiegler B, Kuczynski S, Macartney G, Sung L. Initial development of the Symptom Screening in Pediatrics Tool (SSPedi). Support Care Cancer. 2014 Jan;22(1):71-5. doi: 10.1007/s00520-013-1945-x. Epub 2013 Aug 31. PMID 23995756
- [Background] Molassiotis A, Russell W, Hughes J, Breckons M, Lloyd-Williams M, Richardson J, Hulme C, Brearley S, Campbell M, Garrow A, Ryder W. The effectiveness and cost-effectiveness of acupressure for the control and management of chemotherapy-related acute and delayed nausea: Assessment of Nausea in Chemotherapy Research (ANCHoR), a randomised controlled trial. Health Technol Assess. 2013 Jun;17(26):1-114. doi: 10.3310/hta17260. PMID 23803562